CLINICAL TRIAL: NCT06604533
Title: A Randomized Phase II Trial - Magnetic Resonance Imaging (MRI) Guided Stereotactic Adaptive Radiotherapy for Targeting Abdominal Cancer
Brief Title: Magnetic Resonance Imaging (MRI) Guided Stereotactic Adaptive Radiotherapy for Targeting Abdominal Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Australasian Gastro-Intestinal Trials Group (Network)
Collaborators: Trans Tasman Radiation Oncology Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MR-STAR
Record Dates: First submitted 2024-07-08; First posted 2024-09-19 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-10

CONDITIONS: Abdominal Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: MRI-Linac SABR (Experimental): The treatment planning protocol follows the UK SABR Consortium Guidelines. Patients will be prescribed the maximum isotoxic dose achievable while meeting normal organ tolerances (normal liver, kidney, spinal cord, stomach, duodenum, small and large bowel, heart, lungs, chest wall). The lowest acceptable SABR doses are indicated in the dose range Table within the protocol. The maximum dose/fraction also indicates the maximum the dose can be escalated to for each adaptive session on the MRI-Linac.
  Interventions: Procedure: Intervention: MRI-Linac SABR
- Control: Standard SABR (No Intervention): The treatment planning protocol follows the UK SABR Consortium Guidelines. Patients will be prescribed the maximum isotoxic dose achievable while meeting normal organ tolerances (normal liver, kidney, spinal cord, stomach, duodenum, small and large bowel, heart, lungs, chest wall). The lowest acceptable SABR doses are indicated in the dose range Table within the protocol. The maximum dose/fraction also indicates the maximum the dose can be escalated to for each adaptive session on the MRI-Linac.

INTERVENTIONS:
Procedure: Intervention: MRI-Linac SABR — The treatment planning protocol follows the UK SABR Consortium Guidelines. Patients will be prescribed the maximum isotoxic dose achievable while meeting normal organ tolerances (normal liver, kidney, spinal cord, stomach, duodenum, small and large bowel, heart, lungs, chest wall). The lowest acceptable SABR doses are indicated in the dose range Table within the protocol. The maximum dose/fraction also indicates the maximum the dose can be escalated to for each adaptive session on the MRI-Linac.
  Arms: Intervention: MRI-Linac SABR

SUMMARY:
The aim of this study is to investigate the effect of MRI-guided adaptive stereotactic radiotherapy on local control, survival, and toxicity in the treatment of oligometastatic cancer to the abdomen.

DETAILED DESCRIPTION:
This is an Australian-led multi-centre Phase 2 randomised controlled trial. The aim of this study is to investigate the effect of MRI-guided adaptive stereotactic radiotherapy on LC, survival, and toxicity in the treatment of oligometastatic cancer to the abdomen.

This study will provide one of the first high level phase 2 randomised evidence required to demonstrate this new technology improves patient clinical outcomes and inform the selection of patients for MRI-Linac treatment.

The primary objective is to evaluate the effect of MRI-guided adaptive stereotactic radiotherapy on 2 year LC of treated lesion(s) in patients with abdominal oligometastatic or primary liver cancer.

Aim 1: Quantify the effect of MRI-guided stereotactic radiotherapy on patient outcomes. Patient outcomes will be determined by measuring LC, survival, and safety (toxicity).

Aim 2: Quantify patient dose and cancer targeting accuracy. The ability of MRI-Linacs to treat more patients to a higher dose than standard linacs through adaptive dose-escalation and improved target coverage will be quantified. The delivered dose for each treatment arm will be compared.

Aim 3: Explore functional MRI biomarkers of radiotherapy response prediction. Candidate functional biomarkers of tumour perfusion and diffusion will be identified.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Patients with diagnosis of oligometastatic disease from primary colorectal, upper gastrointestinal (e.g. gastric, oesophagus, pancreatic), breast, non-small cell lung, renal cell, or gynaecological malignancy. Oligometastatic disease with controlled primary disease* and maximum total of 5 metastatic lesions in a maximum of 2 different organ systems in any of the following sites:

  1. Liver
  2. Adrenal
  3. Abdomino-pelvic lymph node
  4. Other abdominal site e.g. pancreatic, renal.
  5. Other pelvic site
  6. Bony or lung is allowed only if in conjunction with an abdominal site above
* De novo or metachronous oligometastatic disease where the original tumour site has been treated with curative intent.

  * Controlled primary disease in metachronous oligometastastic disease defined as at least 3 months since original tumour treated with curative intent and no progression at primary site
  * Controlled primary disease in de novo oligometastatic disease defined as primary tumour site treated with curative intent and no progression at primary site
* Oligometastatic disease: Histological confirmation of primary malignancy (histological confirmation of metastasis is not mandatory but should be performed in any situation where there is any diagnostic uncertainty).
* All oligometastatic sites treatable with SABR.

OR

* Patients with oligo-progressive / oligo-persistent disease in maximum total of 2 oligo-progressive abdominal metastases and in a maximum 2 different organ systems
* Visible imaging defined targets and suitable for treatment with SABR
* Childs Pugh A to B7 (in case of liver treatment)
* ECOG 0 -2
* Patient consented

Exclusion Criteria:

* Contra-indication to MRI
* Previous high dose radiotherapy to a site requiring stereotactic treatment (including SIRTEX). Further SABR treatment of lesions previously treated with SABR or high dose radiotherapy is not permitted in this trial.
* Substantial overlap with a previously treated high dose (definitive or stereotactic dose) radiation volume.
* Primary prostate cancer, carcinoid tumours, germ cell tumours, lymphoma, small cell tumours
* Pregnant women
* Complete response of metastatic disease to systemic therapy (i.e. no target for SABR)
* Competing medical co-morbidity with a more limited prognosis than the cancer diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-07 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Rate of local control (Local Response Rate). | Clinical progress imaging every 3 months post radiotherapy treatment until 3 years post radiotherapy.
  To determine if patients treated with MRI guided stereotactic radiotherapy improves local control. Local control is defined as absence of progression in treated lesion(s) and will be measured via clinical progress imaging (and assessed using RECIST criteria).

CONTACTS AND LOCATIONS:
Overall Officials: Trang Pham, Study Chair — South Western Sydney LHD
Locations (2):
- Australia (2):
  - GenesisCare - St Vincent's Sydney, Darlinghurst, New South Wales
  - Austin Health, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No